CLINICAL TRIAL: NCT06510387
Title: Comparison of Two Bedside Ultrasound Techniques and Standard Methods for Confirmation of Endotracheal Tube Insertion in Intensive Care Patients, A Cross-Sectional Observational Study
Brief Title: Two Bedside Ultrasound Techniques and Standard Methods for Confirmation of Endotracheal Tube Insertion in Intensive Care Patients
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Elsayed Ismaeil Abuharga, Resident of Emergency Medicine and Traumatology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264MS323/9/23
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Two Bedside; Ultrasound; Endotracheal Tube; Intensive Care Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Correct placement group: The research resident will perform ultrasonography using suprasternal and subxiphoid methods to confirm the correct placement of the endotracheal tube.
  Interventions: Device: Ultrasound using suprasternal method; Device: Ultrasound using subxiphoid method
- Incorrect placement group: The research resident will perform ultrasonography using suprasternal and subxiphoid methods.
  Interventions: Device: Ultrasound using suprasternal method; Device: Ultrasound using subxiphoid method

INTERVENTIONS:
Device: Ultrasound using suprasternal method — The research resident will perform suprasternal ultrasound (US) with a curvilinear probe) C6-2) of US machine (Philips Affiniti 50) which will be placed transversely on the suprasternal area just above to the suprasternal notch immediately after intubation, The position of the trachea will be determined by a hyperechoic air-mucosa (A-M) interface with reverberation artifact posteriorly (comet-tail artifact).
  The position of endotracheal tube (ETT), when it is placed in trachea, will be defined as observable contour between A-M and comet-tail artifact. If the second contour appears, it will be similar to the second airway which is called double-tract sign which means that the ETT will be in the esophagus. (7) If the position of the esophagus is suspected of being exactly behind the trachea, operator of ultrasound can specify the location of the esophagus by moving the probe to the left and right sides during scan.
Device: Ultrasound using subxiphoid method — Immediately after suprasternal sonography, the research resident will perform subxiphoid sonography to detect diaphragmatic motion, and information will be recorded.

SUMMARY:
This cross-sectional observational study aims to predict the sensitivity and specificity of ultrasonography using suprasternal and subxiphoid methods to confirm the correct placement of endotracheal tubes compared to standard methods in intensive care patients.

DETAILED DESCRIPTION:
Endotracheal intubation is the primary medical procedure used for securing the airway, confirmation of endotracheal tube (ETT) placement is essential to prevent hypoxia and aspiration. The best primary approach to confirm endotracheal tube placement is observation of the tube passage through the vocal cords followed by assessment based on chest and epigastric auscultation.

Ultrasound machines are now increasingly available in emergency departments and intensive care units. It is a non-invasive, portable and serves as a real-time diagnostic tool with rapid and accurate results.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old.
* Both sex.
* All patients requiring prophylactic airway management e.g (patient with Glasgow Coma Scale <8) with endotracheal intubation in the intensive care unit.

Exclusion Criteria:

* An abnormal airway anatomy.
* Tracheal or endobronchial lesion.
* Significant cervical trauma.
* Cervical abnormality.
* Neck swelling.
* Patients who need cardiopulmonary resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years old, of both sexes undergoing endotracheal intubation admitted to the emergency and traumatology department ICU between October 2023 to September 2024.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy to predict correct placement | 5 minutes after placement of endotracheal tube
  Accuracy in predicting the correct placement of the endotracheal tube will be assessed using Sensitivity and Specificity, positive predictive value (PPV), and negative predictive value (NPV) for each ultrasound technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.